CLINICAL TRIAL: NCT03650894
Title: A Phase II Study of Nivolumab Combined With Bicalutamide and Ipilimumab in Metastatic HER2-negative Breast Cancer
Brief Title: Nivolumab, Ipilimumab, and Bicalutamide in Human Epidermal Growth Factor (HER) 2 Negative Breast Cancer Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Bristol-Myers Squibb (Industry); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-8H3
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Breast Neoplasm Female; Breast Cancer; Breast Carcinoma; Breast Tumor
Keywords: Breast Cancer; Her2 negative breast cancer; Immunotherapy; Opdivo; Nivolumab; Yervoy; Ipilimumab; Bicalutamide; Casodex
MeSH Terms: conditions — Breast Neoplasms | interventions — Nivolumab; Ipilimumab; bicalutamide

STUDY DESIGN:
Intervention Model Description: This is a phase II open-label study of nivolumab combined with ipilimumab and bicalutamide for HER2-negative metastatic or unresectable breast cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab, Ipilimumab, and bicalutamide (Experimental): Participants will receive nivolumab plus ipilimumab combination therapy. Participants should receive nivolumab at a dose of 240 milligrams (mg) fixed dose as a 30-minute intravenous (IV) infusion prepared in 50 milliliter (ml) normal saline (NS) every 2 weeks until progression. Participants should receive ipilimumab at a dose of 1 mg/kilogram as a 30-minute IV infusion prepared in 50 ml NS every 6 weeks. All subjects will take bicalutamide 150mg (3 x 50mg tablets) daily.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: Bicalutamide

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 240 mg IV every 2 weeks
  Other Names: Opdivo
Drug: Ipilimumab — Ipilimumab 1 mg/kg IV every 6 weeks.
  Other Names: Yervoy
Drug: Bicalutamide — Oral bicalutamide 150mg (3 x 50mg tablets) daily
  Other Names: Casodex

SUMMARY:
The goal of this protocol is to evaluate the safety and efficacy of an alternative systemic combination approach that omits or delays the use of chemotherapy in metastatic disease, while improving efficacy and durability of response. The approach combines two potentially effective and previously studied strategies: androgen receptor blockade and immune checkpoint therapy.

DETAILED DESCRIPTION:
This is a phase II trial to assess the clinical efficacy and safety of nivolumab (anti-Programmed Death receptor-1, or anti-PD-1) combined with bicalutamide (Androgen Receptor (AR) inhibitor) and ipilimumab (anti-cytotoxic T-lymphocyte-associated protein 4, or anit-CTLA4) in patients with advanced breast cancer.

This study will include adult women with metastatic or locally advanced unresectable Human Epidermal Growth Factor (HER2)-negative breast cancer (by National Comprehensive Cancer Network (NCCN) criteria). Triple-negative breast cancer tumors will require confirmation of AR positivity at screening. Participants will have had no more than one line of previous chemotherapy in non-curative setting; subjects with metastatic progression within 1 year following completion of curative-intent chemotherapy are eligible if they have not received any additional lines of systemic therapy in the non-curative setting.

Women who meet all of the study inclusion criteria, none of the study exclusion criteria, and agree to participate will receive a combination of the following:

* Intravenous nivolumab 240mg, every 2 weeks until progression or unacceptable toxicity
* Intravenous ipilimumab 1mg/kg, every 6 weeks until progression or unacceptable toxicity
* Oral bicalutamide 150mg, daily until progression or unacceptable toxicity

Participants are to be treated for up to 24 months. Patients who have ongoing response will discontinue ipilimumab and nivolumab after 24 months, but at the discretion of the investigator may continue bicalutamide, and will continue assessments as per standard of care. Any patient who subsequently progresses will have the option to resume treatment upon disease progression.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of 0-1;
* Metastatic or locally advanced unresectable HER2-negative breast cancer (by NCCN criteria);
* Triple Negative Breast Cancer tumors will require confirmation of androgen-receptor (AR) positivity at screening (refer to laboratory manual for guidelines). Local testing permitted for eligibility if reviewed by a designated study pathologist;
* RECIST1.1 measurable disease;
* Participants must be willing (if clinically feasible) to provide a fresh tumor biopsy (or archived tissue). For archived tissue, a tissue block from the most recent biopsy is acceptable if no intervening anti-neoplastic therapies have been administered since the time of biopsy.
* Previous systemic chemotherapy: no greater than one line of previous chemotherapy in non-curative setting; subjects with metastatic progression within 1 year following completion of curative-intent chemotherapy are eligible if they have not received any additional lines of systemic therapy in the non-curative setting.
* Participants must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal patient care.
* Participants must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, tumor biopsies, and other requirements of the study
* Adequate hematologic and liver function (using CTCAE v4). (All baseline laboratory requirements will be assessed and should be obtained within 14 days prior to enrollment): WBC≥2000/μL; Neutrophils≥1500/μL; Platelets≥100 × 103/μL; Hemoglobin ≥9.0 g/dL; AST≤3 × ULN; ALT ≤3 × ULN; Total bilirubin ≤1.5 × ULN (except in participants with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL). Subjects with elevations in LFTs related to underlying hepatic cancer involvement may be considered for enrollment (after discussion with lead PI) if ALT/AST is ≤5 x ULN and Total bilirubin ≤3 × ULN.
* Female and Age ≥18 years. (Men are excluded because of potential confounding effects of sex on correlative analyses)
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study treatment.
* Women must not be breastfeeding
* Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of birth regulation for the duration of treatment with study treatment(s) for a total of 5 months post-treatment completion.

Exclusion Criteria:

* Active brain metastases or leptomeningeal metastases. Participants with brain metastases are eligible if these have been treated and there is no magnetic resonance imaging (MRI except where contraindicated in which CT scan is acceptable) evidence of progression for at least 2 weeks after treatment is complete and within 28 days prior to first dose of study drug administration. Cases must be discussed with the lead PI, Dr. Page. Brain lesions are not considered measurable disease.
* Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, or carcinoma in situ of the cervix. Subjects with prior history of unrelated breast cancer not requiring active therapy may be considered for enrollment, but require discussion with and approval of PI;
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the participant to receive protocol therapy, or interfere with the interpretation of study results.
* Participants must have recovered from the effects of major surgery requiring general anesthetic or significant traumatic injury at least 14 days before enrollment.
* Participants with active, known or suspected autoimmune disease. Participants with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Uncontrolled adrenal insufficiency.
* New York Heart Association (NYHA) Functional Classification of Heart Failure: Class III or Class IV
* All toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue must have resolved to Grade 1 (NCI CTCAE version 4) or baseline before administration of study drug. Participants with toxicities attributed to prior anti-cancer therapy which are not expected to resolve and result in long lasting sequelae, such as peripheral neuropathy grade 2 or less, are permitted to enroll
* Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, or psychiatric illness/social situations that would limit obtaining informed consent or compliance with study requirements.
* Participants who have had a history of acute diverticulitis, intra-abdominal abscess, GI obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation.
* Participants with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity.
* Has known active hepatitis B (e.g. HBsAg reactive) or Hepatitis C (e.g. HCV RNA is detected);
* History of allergy or hypersensitivity to study drug components
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody in the metastatic setting, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways. Previous treatment with anti-PD-1/L1 in the curative setting is allowed if subjects have not received such therapy within one year of screening.
* Prior treatment with bicalutamide, enzalutamide, or any other androgen receptor blocker.
* Use of an investigational agent within 4 weeks of Day 1 visit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females, aged 18 or older
Enrollment: 30 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
iRECIST Clinical Benefit Rate (the number of patients with objective response or ongoing stable disease at week 24 using iRECIST guidelines) | 24 weeks
  To assess the 24-week clinical benefit rate of nivolumab combined with bicalutamide and ipilimumab in advanced HER2-negative breast cancers assessed by radiographic criteria (computed tomography (CT) scan or magnetic resonance imaging (MRI) according to iRECIST criteria.

SECONDARY OUTCOMES:
Assess best overall objective response rate (proportion of patients who achieve a complete or partial response) | 24 months
  Best overall objective response rate will be assessed by radiographic criteria from CT or MRI scans and will be based on RECIST 1.1 and iRECIST criteria
Duration of progression free survival | From first patient enrolled through last patient's progression or 24 months following last patient enrolled, whichever comes first.
  Average length of time between study entry and disease progression or death
Overall survival rate | 24 months.
  Number of patients who are alive

CONTACTS AND LOCATIONS:
Overall Officials: David B. Page, MD, Principal Investigator — Providence Health & Services
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Providence Oncology & Hematology Care Clinic - Eastside, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Providence Cancer Institute — https://oregon.providence.org/our-services/p/providence-cancer-center